CLINICAL TRIAL: NCT01992315
Title: Investigation of Decellularized Adipose Derived-ECM for the Correction of Acquired Soft Tissue Deformities of the Body and Face
Brief Title: Investigation of A-ECM for the Correction of Soft Tissue Defects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aegeria Soft Tissue LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AST Adipose ECM
Record Dates: First submitted 2013-11-14; First posted 2013-11-25 (Estimated); Last update posted 2013-11-25 (Estimated); Status verified 2013-11

CONDITIONS: Disorder of Soft Tissue of Body Wall Region
Keywords: Scar; Soft tissue defect
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adipose-Derived ECM (Experimental)
  Interventions: Device: Adipose-derived ECM

INTERVENTIONS:
Device: Adipose-derived ECM — Each syringe of adipose-derived ECM will hold 2mL and will be for single use only. Up to 3 syringes (6mL total) may be used for each patient. Injections will be made under local anesthesia and sterile conditions using a 23-gauge needle. All injections will be performed in an outpatient clinic setting at study site by the principal investigator who will determine the method, depth, and volume of each implant. Decellularized adipose tissue-derived matrix will be infiltrated into the defect and the underlying musculature as well as the subcutaneous tissue surrounding the defect, with the goal of creating a smooth transition from surrounding structures to the filled defect. This will be performed using a series of multiple punctures or a single puncture with a fanning or threading technique. After the injection is completed, the treatment area will be massaged to conform to the contour of the surrounding tissue and ice will be applied as needed for swelling.

SUMMARY:
Soft tissue injury leads to significant deformity in size, shape and body contour. Adipose tissue, continues to be the tissue of choice in repairing soft tissue defects due to traumatic or other defects. Current autologous fat transfer techniques, however, have a number of limitations including significant donor site morbidity, unpredictable resorption, and the potential for requiring revision. Thus, an "off-the-shelf" material that retains the mechanical and biological properties of adipose tissue would be ideal for the reconstruction.

Extracellular matrix (ECM)-based biomaterials have the potential to be a non-immunogenic biological scaffold for adipose tissue engineering for repair of soft tissue defects. Our collaborators have recently generated a novel tissue-derived material to improve soft tissue reconstruction. The final, processed adipose tissue does not contain cellular components, yet retains the native architecture and bioactivity of the original adipose tissue. The tissue is then further processed into particles to create an injectable implant. In preclinical models, we have demonstrated that human adipose tissue can be decellularized by mechanical processing with preservation of matrix ultrastructure. Histologic analysis two-weeks after implantation into rats showed minimal inflammatory reaction and good tissue integration of the decellularized, dilipidized, adipose derived-ECM.

The goal of the study is to 1) evaluate the safety and compatibility of the soft tissue implant, and 2) determine the efficacy of this ECM replacement in soft tissue injuries after 6 weeks. Specifically, the volume of the soft tissue defect will be determined before implantation and at multiple time points over the following 6 weeks. We hypothesize that the decellularized adipose ECM will retain at least 50% volume and surface area after 6 weeks. If our results are promising, decellularized adipose derived-ECM may be a viable alternative to autologous tissue transplantation for correction of soft tissue deformity.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, ages 20-50, with previous congenital or acquired soft tissue deformities of the body or face that are willing to have photographs taken may join this study

Exclusion Criteria:

* pregnant women, patients with known immunocompromise or wound healing disorders

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2014-03; Primary Completion 2015-06 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Clinical assessment of toxicity associated with soft tissue injection of Adipose-derived ECM | 6 weeks
  At each post-injection visit, week 1, 4, and 6, the principal investigator will examine patients for presence of adverse events such as toxicity, pain/inflammation at the site of injection

SECONDARY OUTCOMES:
Objective assessment of volume retention following soft tissue injection of Adipose-derived ECM | 6 weeks
  At each visit, week 1, 4, and 6, 3-D photography will be performed to assess volume retention

OTHER OUTCOMES:
Measure of physician satisfaction | 6 weeks
  Physician satisfaction will after using the decellularized adipose derived-ECM. This will be performed using a questionnaire to be completed by participating physicians.
Measure of participant satisfaction | 6 weeks
  Participant satisfaction measurement will be performed using a survey to completed by participants at each follow up visit, week 1, 4 and 6.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Lickstein, MD, Principal Investigator — Cosmetic Surgery Center of Maryland
Locations (1):
- Cosmetic Surgery Center of Maryland, Towson, Maryland, United States

REFERENCES:
- [Background] Wu I, Nahas Z, Kimmerling KA, Rosson GD, Elisseeff JH. An injectable adipose matrix for soft-tissue reconstruction. Plast Reconstr Surg. 2012 Jun;129(6):1247-1257. doi: 10.1097/PRS.0b013e31824ec3dc. PMID 22327888